CLINICAL TRIAL: NCT00232401
Title: The Circadian Rhythm of Urine Output in Healthy Infants
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Birgitte Mahler, Aarhus University hospital
Organization: University of Aarhus (Other)
Other Study IDs: Neo.02.2005
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: urine; circadian rhythm

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to describe the 24-hour urine output including the urinary excretion of hormones, electrolytes and other osmotically active substances in healthy children age 0 to 3 years old.

DETAILED DESCRIPTION:
The purpose of this study is to describe the 24-hour urine output including the urinary excretion of hormones, electrolytes and other osmotically active substances in healthy children age 0 to 3 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, free of medication

Exclusion Criteria:

* History of urinary diseases

Ages: 6 Days to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2005-10; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Mahler, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University, Aarhus, Denmark